CLINICAL TRIAL: NCT00110396
Title: A Multicentre, Single Arm, Open-Label, Phase IIIB Study to Evaluate the Safety and Antigenicity of Rebif® (Interferon-beta-1a) in Subjects With Relapsing Forms of Multiple Sclerosis
Brief Title: Rebif New Formulation (RNF) in Relapsing Forms of Multiple Sclerosis
Acronym: RNF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Susan Fischer, EMD Serono Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25632
Record Dates: First submitted 2005-05-06; First posted 2005-05-09 (Estimated); Results first posted 2010-07-09 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Relapsing forms of multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

ARMS (1):
- Rebif New Formulation Cohort (Experimental)
  Interventions: Biological: Interferon-beta-1a FBS-free/HSA-free

INTERVENTIONS:
Biological: Interferon-beta-1a FBS-free/HSA-free — Pre-filled syringes 44mcg/injected subcutaneous 3x per week. Total study period is 96 weeks.

SUMMARY:
The primary objective of the study is to compare the immunogenicity of the new fetal bovine serum (FBS)-free/human serum albumin (HSA)-free Rebif® formulation (RNF) to historical data.

DETAILED DESCRIPTION:
As has been seen with other recombinant protein molecules, the use of injectable recombinant proteins may result in the development of neutralising antibodies (NAbs). Antibodies are considered neutralising by their ability to inhibit the biological effect of interferon in a bioassay system. EMD Serono has actively pursued improvements in the formulation of interferon (IFN) beta-1a to reduce aggregate levels and to develop a formulation that is HSA-free. Reducing aggregates should reduce antigenicity of the product while removal of HSA may have an unpredictable effect on antigenicity. EMD Serono will conduct a study to assess the immunogenicity and safety of the new HSA-free formulation, manufactured using IFN-ß-1a drug substance produced by a new clone from the FBS-free process.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a relapsing form of Multiple Sclerosis (MS); diagnosis of MS is in accordance with the McDonald criteria
* Participant is eligible for interferon therapy
* Participant is between 18 and 60 years old
* Participant has an Expanded Disability Status Scale (EDSS) < 6.0.
* Participant is willing to follow study procedures
* Participant has given written informed consent
* Female participants must be neither pregnant nor breast-feeding, and must lack childbearing potential, as defined by either:
* Being post-menopausal or surgically sterile, or
* Using a hormonal contraceptive, intra-uterine device, diaphragm with spermicide or condom with spermicide for the duration of the study.
* Confirmation that the participant is not pregnant must be established by a negative serum or urinary hCG test within 7 days prior to start of study treatment. A pregnancy test is not required if the participant is post-menopausal or surgically sterile.

Exclusion Criteria:

* Participant has a Clinically Isolated Syndrome (CIS), Primary Progressive MS, or Secondary Progressive MS without superimposed relapses.
* Participant had any prior interferon beta therapy (either beta-1b or beta-1a)
* Participant has an ongoing MS relapse.
* Participant received any other approved disease modifying therapy for MS (e.g. glatiramer acetate) or any cytokine or anti-cytokine therapy within the 3 months prior to Study Day 1(SD1).
* Participant had prior use of cladribine or has previously received total lymphoid irradiation.
* Participant received oral or systemic corticosteroids or adrenocorticotropic hormone (ACTH) within 30 days of SD1.
* Participant received intravenous immunoglobulins or underwent plasmapheresis within the 6 months prior to SD1.
* Participant received immunomodulatory or immunosuppressive therapy (including but not limited to cyclophosphamide, cyclosporin, methotrexate, azathioprine, linomide, mitoxantrone, teriflunomide, natalizumab, laquinimod, Campath) within the 12 months prior to SD1.
* Participant requires chronic or monthly pulse corticosteroids during the study.
* Participant received any investigational drug or experimental procedure within 12 weeks of SD1.
* Participant has inadequate liver function, defined by a total bilirubin, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or alkaline phosphatase > 2.5 times the upper limit of the normal values.
* Participant has inadequate bone marrow reserve, defined as a white blood cell count less than 0.5 x lower limit of normal.
* Participant suffers from current autoimmune disease.
* Participant suffers from major medical or psychiatric illness that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the study protocol.
* Participant has a known allergy to IFN or the excipients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2005-01; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Stubinski, MD, Study Director — Merck Serono SA - Geneva
Locations (1):
- Local US Medical Information, Rockland, Massachusetts, United States

REFERENCES:
- [Result] Giovannoni G, Barbarash O, Casset-Semanaz F, Jaber A, King J, Metz L, Pardo G, Simsarian J, Sorensen PS, Stubinski B; RNF Study Group. Immunogenicity and tolerability of an investigational formulation of interferon-beta1a: 24- and 48-week interim analyses of a 2-year, single-arm, historically controlled, phase IIIb study in adults with multiple sclerosis. Clin Ther. 2007 Jun;29(6):1128-45. doi: 10.1016/j.clinthera.2007.06.002. PMID 17692727
- [Result] Giovannoni G, Barbarash O, Casset-Semanaz F, King J, Metz L, Pardo G, Simsarian J, Sorensen PS, Stubinski B; Rebif New Formulation Study Group. Safety and immunogenicity of a new formulation of interferon beta-1a (Rebif New Formulation) in a Phase IIIb study in patients with relapsing multiple sclerosis: 96-week results. Mult Scler. 2009 Feb;15(2):219-28. doi: 10.1177/1352458508097299. Epub 2008 Aug 28. PMID 18755819
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 25 Jan 2005 and attended the last visit on 16 April 2007. Two hundred and eighty two participants were screened for enrollment and 260 were enrolled.
Pre-assignment Details: Screening phase of up to 28 days before the start of interferon-beta-1a treatment. There were 47 centres in: Argentina (5), Australia (4),Canada (1), Denmark (1),Ireland (2), Israel (2), Lithuania(2), Russia (10), Spain (4), Sweden (1), UK (5) and US (10). 1 additional centre in Australia screened 1 participant who was not enrolled into the trial.
Groups:
- Rebif New Formulation (RNF) Cohort: Interferon-beta-1a FBS-free/HSA-free Pre-filled syringes 44mcg/injected subcutaneous 3x per week
Period: Overall Study
Arm/Group | Rebif New Formulation (RNF) Cohort
Started | 260
Completed | 224 (260 participants included in the Safety Population.207 completed treatment. 224 completed the trial)
Not Completed | 36
Not completed — Adverse Event | 15
Not completed — Lost to Follow-up | 1
Not completed — Administration of plasmapheresis | 1
Not completed — Initiated mitoxantrone therapy | 1
Not completed — Lack of Efficacy | 1
Not completed — Decided not to continue treatment | 1
Not completed — Patient non-compliance | 1
Not completed — Patient refused to continue | 1
Not completed — Patient refused to participate | 1
Not completed — Patient will | 1
Not completed — Patient's decision | 1
Not completed — Participation in MS vaccine study | 1
Not completed — Pregnancy | 1
Not completed — Pregnancy (Protocol violation) | 2
Not completed — Protocol Violation | 2
Not completed — Patient refused to come back | 1
Not completed — The patient has refused | 2
Not completed — The patient has refused to visit site | 1
Not completed — Patient is to be administered copaxone | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rebif New Formulation (RNF) Cohort
Number analyzed (Participants) | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 260
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186
  Male | 74
Region of Enrollment [Number; unit: participants]
  Argentina | 14
  Australia | 10
  Canada | 4
  Denmark | 4
  Ireland | 4
  Israel | 4
  Lithuania | 20
  Russian Federation | 134
  Spain | 13
  Sweden | 5
  United Kingdom | 23
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Neutralising Antibody (NAb) Positive at the Week 96 Visit.
Description: The NAb positive value was defined as NAb value greater or equal to 20 NU/mL. NAbs were detected using a viral cytopathic assay.
Time Frame: 96 weeks
Population: ITT (One participant did not have any post-baseline NAb assessments). LOCF imputation
Measure: Number; unit: participants
Arm/Group | Rebif New Formulation (RNF) Cohort
Number analyzed (Participants) | 259
participants | 45

2. Secondary Outcome: Number of Participants Who Were Neutralising Antibody (NAb) Positive at Anytime During the Study
Description: as for outcome 1
Time Frame: 96 weeks
Population: ITT (One participant did not have any post-baseline NAb assessments). LOCF imputation
Measure: Number; unit: participants
Arm/Group | Rebif New Formulation (RNF) Cohort
Number analyzed (Participants) | 259
participants | 49

3. Secondary Outcome: Number of Participants With Binding Antibodies (BAb) at Week 96
Description: Presence of BAbs. BAbs were measured by ELISA (Enzyme-linked immunosorbent assay).
Time Frame: 96 weeks
Population: ITT (One participant did not have any post-baseline NAb assessments) LOCF imputation
Measure: Number; unit: Participants
Arm/Group | Rebif New Formulation (RNF) Cohort
Number analyzed (Participants) | 259
Participants | 74

ADVERSE EVENTS:
Time Frame: Adverse event reporting began at signature of informed consent and continued until 4 weeks after the last administration of trial medication.
Description: Investigator recorded AE's at every visit.
Arm/Group | Rebif New Formulation (RNF) Cohort
Serious Adverse Events (participants affected / at risk) | 15/260
Other Adverse Events (participants affected / at risk) | 247/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rebif New Formulation (RNF) Cohort (N=260)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 1 (1)
Depression (Psychiatric disorders) | 3 (3)
Hypomania (Psychiatric disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 1 (1)
Periproctitis (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rebif New Formulation (RNF) Cohort (N=260)
Influenza like illness (General disorders) | 176 (329)
Headache (Nervous system disorders) | 98 (229)
Injection site erythema (General disorders) | 63 (76)
Nausea (Gastrointestinal disorders) | 26 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (31)
Injection site haemorrhage (General disorders) | 25 (30)
Fatigue (General disorders) | 24 (26)
Upper respiratory tract infection (Infections and infestations) | 23 (36)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (32)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 (26)
Alanine aminotransferase increased (Investigations) | 19 (22)
Dizziness (Nervous system disorders) | 19 (22)
Pyrexia (General disorders) | 18 (32)
Chills (General disorders) | 18 (24)
Neutropenia (Blood and lymphatic system disorders) | 18 (23)
Nasopharyngitis (Infections and infestations) | 17 (22)
Diarrhoea (Gastrointestinal disorders) | 17 (21)
Injection site pain (General disorders) | 17 (21)
Asthenia (General disorders) | 16 (25)
Viral upper respiratory tract infection (Infections and infestations) | 15 (25)
Aspartate aminotransferase increased (Investigations) | 15 (19)
Urinary tract infection (Infections and infestations) | 14 (27)
Vomiting (Gastrointestinal disorders) | 13 (16)
Insomnia (Psychiatric disorders) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SPONSOR shall have the right to publish or present any results or information, including the Study Results, arising in connection with the STUDY for any purposes. The INSTITUTION, its officers, agents, employees and affiliated entities shall not publish or use any results or information arising in connection with the STUDY, including the Study Results, for professional, research, training or other purposes without SPONSOR's prior written consent.